CLINICAL TRIAL: NCT03702010
Title: Randomized, Single-blind, Multicenter, Crossover, Controlled Clinical Trial to Compare Difference on the Visual Analogue Scale With Two Modes of Spinal Cord Stimulation in Patients With Post-Laminectomy Syndrome in Testing Phase
Brief Title: Spinal Cord Stimulation in Patients With Post-Laminectomy Syndrome in Testing Phase
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundación Instituto de Estudios de Ciencias de la Salud de Castilla y León (Other)
Collaborators: Instituto de Investigación Biomédica de Salamanca (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Health Services Research
Other Study IDs: EST-MED-2018-01; E.C.P.S. 18/1398 (Other: IBSAL (INSTITUTO DE INVESTIGACIÓN BIOMÉDICA DE SALAMANCA))
Record Dates: First submitted 2018-09-25; First posted 2018-10-10 (Actual); Results first posted 2021-09-01 (Actual); Last update posted 2021-09-01 (Actual); Status verified 2021-08

CONDITIONS: Laminectomy; Post-laminectomy Syndrome; Spinal Cord Syndrome; Failed Back Surgery Syndrome
Keywords: Spinal cord stimulation; Back surgery; Chronic pain
MeSH Terms: conditions — post laminectomy syndrome; Spinal Cord Injuries; Failed Back Surgery Syndrome; Chronic Pain

STUDY DESIGN:
Intervention Model Description: Single-blind, multicenter, crossover
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CME branch (Active Comparator): In this study, the conventional spinal cord stimulation method (control Branch-CME branch)
  Interventions: Device: spinal cord stimulation conventional
- EME branch (Experimental): In this study, the experimental spinal cord stimulation method are used in the same patient with the EVOLVE programming guide (EME branch)
  Interventions: Device: spinal cord stimulation experimental

INTERVENTIONS:
Device: spinal cord stimulation conventional — If the patient has been assigned to the branch of the CME control group, after mapping the search for the pain zone, the neurostimulator is programmed to conventional stimulation.
  Other Names: CME
  Arms: CME branch
Device: spinal cord stimulation experimental — If the patient has been randomized to the branch of the EME experimental group, after a mapping of the search for the pain zone, a 90% subthreshold stimulation is programmed.
  Other Names: EME
  Arms: EME branch

SUMMARY:
Traditionally, pain relief through spinal cord stimulation has been associated with the appearance of paresthesia in the affected area. Several parameters are set to maximize the overexposure zone, such as frequency,and pulse width. Although this technique has improved pain in many patients, paresthesia itself can be uncomfortable. Traditionally, the occurrence of paresthesias has been considered to be a predictor of success in pain elimination, while the non-occurrence of paresthesias would indicate failure. So far, few studies have reported pain relief below the threshold of onset of paresthesia. Some clinical trials for pathologies other than the one considered in this study have achieved relief below the threshold by reducing the amplitude of the stimulus. Recently, however, it has been observed in a pilot study that, by increasing the frequency of spinal cord stimulation to 1 kilohertz, it is possible to significantly improve pain relief compared to less frequent conventional stimulation based on the occurrence of paresthesias.

A recent review by the Cochrane Library concluded that conventional spinal cord stimulation for pain relief of Failed Back Surgery Syndrome (or FBSS) requires further clinical studies and better designs to demonstrate its superiority over other therapeutic options. Therefore, although spinal cord stimulation is accepted by the Food and Drug Administration (FDA) and the European Medicines Agency (EMA), new techniques are being introduced that offer better results in terms of pain relief. Among these techniques, there is the high frequency mode, which allows avoiding the annoying sensation of paresthesia that substitutes pain with the conventional technique. In order to provide greater rigour and scientific quality, the present study is proposed, in which the conventional spinal cord stimulation (CME) technique (control branch or CME) is compared with paresthesias and a standard frequency (60 hertz) with a high frequency (1000 hertz) EVOLVE system (Evolve workflow - standardized guidance to simplify the trial and implant experience and optimize patient outcomes) (experimental branch or EME) by means of a design with a high degree of scientific evidence, randomising the global sample of patients to each of the two branches of stimulation in the study (blind to the patient) and crossing the branches after a period of washing

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years of age.
* Patients with FBSS syndrome with leg pain or leg and back pain.
* Get a score on the visual analogue scale (VAS) ≥ 7.
* Have received medical pharmacological treatment for at least 6 months after back surgery.
* The patient has signed the informed consent form.

Exclusion Criteria:

* Patients under 18 years of age.
* Patients who require a diathermic energy source (microwave, ultrasound or short wave).
* Patients with a pacemaker.
* Patients carrying a defibrillator.
* Patient with a cochlear implant.
* Patients with other active implanted devices.
* Patients who are scheduled to have any of the following procedures during the study period: an MRI, defibrillation or cardioversion, electrocautery, lithotripsy, radiofrequency or microwave ablation, and any other high-frequency ultrasound procedure,
* Women of childbearing age who do not use adequate contraception.
* Pregnant or breastfeeding.
* Participation in another trial.
* Patients who have expressed a desire not to participate in the study and have not formed informed consent.
* Patients with a failed spinal cord stimulation implant previously

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2018-11-20 (Actual); Primary Completion 2020-07-01 (Actual); Study Completion 2020-07-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Francisco J Sánchez-Montero, MD, Study Director — IBSAL-Instituto de Investigación Biomédica de Salamanca
Locations (2):
- Spain (2):
  - Hospital San Pedro de Logroño, Logroño, La Rioja
  - Complejo Asistencial Universitario de Salamanca, Salamanca

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Planned enrollment: 24. Final enrollment: 27. Screened: 28.
Pre-assignment Details: 27 of 28 patients screened were randomized, as one patient did not meet inclusion/exclusion criteria.
  All patients underwent both treatments, as the study design was cross-section.
Groups:
- CME - EME Branch: In this study, the conventional spinal cord stimulation method (control Branch-CME branch)
  CME control group: after mapping the search for the pain area, the neurostimulator is programmed to conventional stimulation with paresthesia at 60 Hz and a pulse width between 300-450 μs, for 5 days.
  The device is then deprogrammed and a 2-day washout period is initiated.
  On day 7, EME protocol is initiated: stimulation is programmed at 90% of the subthreshold with a pulse width of 90 μs and frequency of 1000 Hz, placing the bipole in the T9-T10 space, for 5 days.
- EME - CME Branch: In this study, the experimental spinal cord stimulation method are used in the same patient with the EVOLVE programming guide (EME branch)
  EME experimental group: fter mapping the search for the pain area, the neurostimulator is programmed at 90% of the subthreshold with a pulse width of 90 μs and frequency of 1000 Hz, placing the bipole in the T9-T10 space, for 5 days.
  The device is then deprogrammed and a 2-day washout period is initiated.
  On day 7, conventional CME stimulation is programmed with paresthesia at 60 Hz and a pulse width between 300-450 μs, for 5 days.
Period: First Stimulation (5 Days)
Arm/Group | CME - EME Branch | EME - CME Branch
Started | 13 | 14
Completed | 13 | 14
Not Completed | 0 | 0
Period: Washout + Second Stimulation (2+5days)
Arm/Group | CME - EME Branch | EME - CME Branch
Started | 13 | 14
Completed | 13 | 14
Not Completed | 0 | 0
Period: Follow-up (30days)
Arm/Group | CME - EME Branch | EME - CME Branch
Started | 13 | 14
Completed | 11 | 12
Not Completed | 2 | 2
Not completed — Lack of Efficacy | 2 | 2

BASELINE CHARACTERISTICS:
Population: All participants underwent both neurostimulation protocols, as it was a crossover study.
Groups:
- CME - EME Branch: After mapping the search for the pain area, the neurostimulator is programmed to conventional stimulation (CME) with paresthesia at 60 Hz and a pulse width between 300-450 μs, for 5 days.
  The device is then deprogrammed and a 2-day washout period is initiated.
  On day 7, EME experimental protocol is initiated: stimulation is programmed at 90% of the subthreshold with a pulse width of 90 μs and frequency of 1000 Hz, placing the bipole in the T9-T10 space, for 5 days.
- EME - CME Branch: After mapping the search for the pain area, the neurostimulator is programmed to EME experimental protocol is initiated: stimulation is programmed at 90% of the subthreshold with a pulse width of 90 μs and frequency of 1000 Hz, placing the bipole in the T9-T10 space, for 5 days.
  The device is then deprogrammed and a 2-day washout period is initiated.
  On day 7, conventional stimulation (CME) stimulation is programmed with paresthesia at 60 Hz and a pulse width between 300-450 μs, for 5 days.
- Total: Total of all reporting groups
Arm/Group | CME - EME Branch | EME - CME Branch | Total
Number analyzed (Participants) | 13 | 14 | 27
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.8 (13.1) | 53.9 (12.6) | 52.4 (12.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 4 | 10
  Male | 7 | 10 | 17
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Spain | 13 | 14 | 27
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m2] | 26.0 (4.3) | 28.2 (4.3) | 27.2 (4.4)

OUTCOME MEASURES:

1. Primary Outcome: Comparing Visual Analogue Scale (VAS)
Description: Visual analogue scale (VAS) at the end of each test phase (either with conventional spinal cord stimulation or with EVOLVE). VAS consists of a 10 centimeter (cm) line, whose ends are defined as the extreme limits of pain (left end corresponds with the absence of pain and the right end with the maximum amount of pain).
  The patient is asked to point out in the line the place that better correspond to his/her pain, ranging from 0 to 10.
Time Frame: Baseline, After first stimulation (5days), after washout and second stimulation (12 days), After 30-day follow-up (42 days)
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- CME -EME Branch: Conventional CME: after mapping the search for the pain area, the neurostimulator is programmed to conventional stimulation with paresthesia at 60 Hz and a pulse width between 300-450 μs, for 5 days.
  The device is then deprogrammed and a 2-day washout period is initiated.
  On day 7, EME protocol is initiated: stimulation is programmed at 90% of the subthreshold with a pulse width of 90 μs and frequency of 1000 Hz, placing the bipole in the T9-T10 space, for 5 days.
- EME-CME Branch: EVOLVE programming guide (EME): after mapping the search for the pain area, the neurostimulator is programmed at 90% of the subthreshold with a pulse width of 90 μs and frequency of 1000 Hz, placing the bipole in the T9-T10 space, for 5 days
  The device is then deprogrammed and a 2-day washout period is initiated.
  On day 7, CME protocol is initiated: stimulation is programmed to conventional stimulation with paresthesia at 60 Hz and a pulse width between 300-450 μs, for 5 days.
Arm/Group | CME -EME Branch | EME-CME Branch
Number analyzed (Participants) | 13 | 14
score on a scale
  Baseline | 9.3 (1.1) | 8.6 (1.0)
  After first stimulation (day +5) | 5.7 (1.7) | 4.9 (2.3)
  After washout and second stimulation (day +12) | 5.5 (2.2) | 5.2 (2.4)
  After Follow-up (day +42) | 4.6 (1.8) | 4.2 (2.2)
Statistical Analysis 1: Comparison: CME -EME Branch vs EME-CME Branch; Baseline VAS; Test type: Superiority; p = 0.112, t-test, 2 sided
Statistical Analysis 2: Comparison: CME -EME Branch vs EME-CME Branch; After first stimulation VAS; Test type: Superiority; p = 0.323, t-test, 2 sided
Statistical Analysis 3: Comparison: CME -EME Branch vs EME-CME Branch; After second stimulation; Test type: Superiority; p = 0.760, t-test, 2 sided
Statistical Analysis 4: Comparison: CME -EME Branch vs EME-CME Branch; End of Follow-up; Test type: Superiority; p = 0.624, t-test, 2 sided

2. Secondary Outcome: Change (%) in VAS Scale at the End of Treatment.
Description: Change (%) in Visual Analogue Scale (VAS) at the end of treatment.
  * Δ = [(VAS Initial Visit - VAS Final Visit) / VAS initial visit] *100
  Please note that positive values indicate a decrease in the VAS scale, which would indicate pain relief, as it was calculated as the value at the earlier time point minus the value at the later time point.
Time Frame: After first stimulation (Five days after baseline), After second stimulation (12 days after baseline), at the end of follow-up (42 days after baseline)
Measure: Mean (Standard Deviation); unit: percentage of VAS change
Groups:
- CME - EME Branch: Conventional spinal cord stimulation (CME) method for 5 days. Washout of 2 days. Experimental spinal cord stimulation (EME) for 5 days.
- EME - CME Branch: Experimental spinal cord stimulation (EME) method for 5 days. Washout of 2 days. Conventional spinal cord stimulation (CME) for 5 days.
Arm/Group | CME - EME Branch | EME - CME Branch
Number analyzed (Participants) | 13 | 14
percentage of VAS change
  After first stimulation | 42.4 (26.0) | 37.4 (20.6)
  After second stimulation | 37.8 (29.1) | 41.5 (20.3)
  End of follow-up | 50.1 (28.1) | 48.8 (21.5)
Statistical Analysis 1: Comparison: CME - EME Branch vs EME - CME Branch; After first stimulation; Test type: Superiority; p = 0.589, t-test, 2 sided
Statistical Analysis 2: Comparison: CME - EME Branch vs EME - CME Branch; After second stimulation; Test type: Superiority; p = 0.704, t-test, 2 sided
Statistical Analysis 3: Comparison: CME - EME Branch vs EME - CME Branch; End of Follow-up; Test type: Superiority; p = 0.908, t-test, 2 sided

3. Secondary Outcome: Evaluation Disability
Description: Oswestry Disability Index of the patients: it is a questionnaire consisting of 10 questions with 6 possible answers each. Every answer gives a punctuation from 0 (less disability) to 5 (more disability).
  This scale is expressed in percentage in which 0 percentage (%) would the least disability and 100 percentage (%) would represent the maximum disability.
Time Frame: Baseline, After first stimulation (+5 days), After washout and second stimulation (+12 days), at the end of follow-up (+42days)
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- CME - EME Branch: CME conventional stimulation for 5 days, Washout for 2 days. EME evolve experimental stimulation for 5 days.
- EME - CME Branch: EVOLVE programming guide (EME) experimental stimulation for 5 days. Washout for 2 days. Conventional stimulation (CME) for 5 days.
Arm/Group | CME - EME Branch | EME - CME Branch
Number analyzed (Participants) | 13 | 14
score on a scale
  Baseline | 59.8 (14.1) | 65.7 (10.5)
  After first stimulation | 44.7 (15.8) | 41.5 (21.4)
  After second stimulation | 43.7 (18.7) | 43.7 (21.8)
  End of Follow-up | 21.8 (21.6) | 24.9 (15.4)
Statistical Analysis 1: Comparison: CME - EME Branch vs EME - CME Branch; Baseline; Test type: Superiority; p = 0.231, t-test, 2 sided
Statistical Analysis 2: Comparison: CME - EME Branch vs EME - CME Branch; After first stimulation; Test type: Superiority; p = 0.663, t-test, 2 sided
Statistical Analysis 3: Comparison: CME - EME Branch vs EME - CME Branch; After second stimulation; Test type: Superiority; p = 0.998, t-test, 2 sided
Statistical Analysis 4: Comparison: CME - EME Branch vs EME - CME Branch; End of Follow-up; Test type: Superiority; p = 0.713, t-test, 2 sided

4. Secondary Outcome: Number of Participants With Adverse Events in Each Arm
Description: Considering as an adverse event those that result in death, or in severe harm to patient's health (lesion that threatens life, permanent harm on an organ or corporal function, or process that needs a medical or surgical intervention to avoid permanent harm)
Time Frame: 42 days from baseline
Measure: Count of Participants; unit: Participants
Groups:
- CME - EME: Conventional stimulation for 5 days Washout for days Experimental stimulation for 5 days
- EME - CME: EVOLVE stimulation for 5 days Washout for 2 days Conventional stimulation for 5 days.
Arm/Group | CME - EME | EME - CME
Number analyzed (Participants) | 13 | 14
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: From baseline to the end of Follow-up (42 days).
Groups:
- CME - Conventional Stimulation: Conventional stimulation with paresthesia at 60 Hz and a pulse width between 300-450 μs, for 5 days.
- EME - EVOLVE Experimental Stimulation: The neurostimulator is programmed to stimulation is programmed at 90% of the subthreshold with a pulse width of 90 μs and frequency of 1000 Hz, placing the bipole in the T9-T10 space, for 5 days.
Arm/Group | CME - Conventional Stimulation | EME - EVOLVE Experimental Stimulation
All-Cause Mortality (participants affected / at risk) | 0/27 | 0/27
Serious Adverse Events (participants affected / at risk) | 0/27 | 0/27
Other Adverse Events (participants affected / at risk) | 3/27 | 4/27
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CME - Conventional Stimulation (N=27) | EME - EVOLVE Experimental Stimulation (N=27)
Pain (Surgical and medical procedures) | 0 (0) | 1 (1) — One patient reported pain in the surgical wound, and also experienced abnormal stimulation.
Electrode migration (Surgical and medical procedures) | 1 (1) | 2 (2)
post-dural puncture headache (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) — two dural punctures resulting in post-dural puncture headache (one episode on each branch)
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Abnormal stimulation (Surgical and medical procedures) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-06-04): https://cdn.clinicaltrials.gov/large-docs/10/NCT03702010/Prot_SAP_000.pdf
  • Informed Consent Form (2018-05-08): https://cdn.clinicaltrials.gov/large-docs/10/NCT03702010/ICF_001.pdf